CLINICAL TRIAL: NCT05942638
Title: Longitudinal Assessment of Post-concussion Driving in Young Adults
Acronym: LAPDYA
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Georgia (Other)
Collaborators: Emory University (Other); University of Kansas (Other); Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Julianne Schmidt, Associate Professor, University of Georgia
Other Study IDs: PROJECT00007249
Record Dates: First submitted 2023-04-28; First posted 2023-07-12 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Brain Injuries, Traumatic; Concussion, Brain; Brain Injury Traumatic Mild
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussion Group
- Control Group

SUMMARY:
Upwards of 3.8 million concussions occur annually in the United States. Driving is a highly complicated activity that requires visual, motor, and cognitive skills, which are commonly impaired after concussion. Yet, the time course of post-concussion driving impairment has not been characterized. There is a critical need to 1) determine when concussed individuals should return to driving and 2) identify the key concussion assessment predictors of readiness to return to driving. In the absence of formal recommendations, impaired concussed drivers are at risk to themselves and others on the road.

The first specific aim is to compare simulated driving between concussed individuals and non-concussed yoked matched controls across five longitudinal timepoints (pre-injury baseline, day 2, day 4, asymptomatic, and unrestricted medical clearance) and daily naturalistic driving from day 2 to day 9.

Driving recommendations must be appropriate and necessitated by concussion impairments, since excessively strict recommendations wrongfully strip concussed patients of their independence and may dissuade individuals from seeking medical care. The second specific aim is to identify widely used concussion assessment outcomes that predict simulated driving performance among concussed individuals throughout concussion recovery.

To address these aims, 100 concussed and 100 yoked matched control young adult college athletes will complete a simulated driving assessment and a robust concussion assessment battery at pre-injury baseline, day 2, day 4, asymptomatic, and unrestricted medical clearance. Naturalistic driving (measured with in-car global positioning systems) will be captured from day 2 to day 9 (7 days total).

This study will determine the acute and subacute time course of post-concussion driving impairment and determine key predictors of post-concussion driving performance. Results from this innovative approach will have a broad and positive impact that will improve the safety of both concussed individuals and the general population, guide the practices of health professionals, inform the future work of researchers, and substantiate the work of policy-makers by providing evidence-based recommendations for managing post-concussion driving.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Possesses a valid driver's license
* 1 year or more of driving experience
* Normal or corrected-to-normal vision
* Rostered on an organized athletic team at the college level
* (Concussion Group Only) Diagnosed with concussion by a physician and meet inclusion criteria above.

Exclusion Criteria:

* Four or more previous concussions
* A concussion within the past 6 months
* History of any major neurological disorders or injuries
* Current use of any medications that evoke drowsiness (prescription or over the counter)
* Current orthopedic condition that interferes with driving (e.g. a walking boot, shoulder immobilizer)
* Heavy use of alcohol (binge drinking 5+ days in the past 30 days)
* Any illegal drug use (any illegal substance use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Athletes rostered in an organized sport at the collegiate level
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Centerline Crossings (count) | Pre-injury baseline
  Count of centerline crossings during a custom STISIM3 driving simulation scenario
Centerline Crossings (count) | Day 2
  Count of centerline crossings during a custom STISIM3 driving simulation scenario
Centerline Crossings (count) | Day 4
  Count of centerline crossings during a custom STISIM3 driving simulation scenario
Centerline Crossings (count) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Count of centerline crossings during a custom STISIM3 driving simulation scenario
Centerline Crossings (count) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Count of centerline crossings during a custom STISIM3 driving simulation scenario
Road edge excursions (count) | Pre-injury baseline
  Count of road edge excursions during a custom STISIM3 driving simulation scenario
Road edge excursions (count) | Day 2
  Count of road edge excursions during a custom STISIM3 driving simulation scenario
Road edge excursions (count) | Day 4
  Count of road edge excursions during a custom STISIM3 driving simulation scenario
Road edge excursions (count) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Count of road edge excursions during a custom STISIM3 driving simulation scenario
Road edge excursions (count) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Count of road edge excursions during a custom STISIM3 driving simulation scenario
Total Collisions (count) | Pre-injury baseline
  Count of collisions during a custom STISIM3 driving simulation scenario
Total Collisions (count) | Day 2
  Count of collisions during a custom STISIM3 driving simulation scenario
Total Collisions (count) | Day 4
  Count of collisions during a custom STISIM3 driving simulation scenario
Total Collisions (count) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Count of collisions during a custom STISIM3 driving simulation scenario
Total Collisions (count) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Count of collisions during a custom STISIM3 driving simulation scenario
Standard Deviation of Lane Position (feet) | Pre-injury baseline
  Variability of lateral lane position during a custom STISIM3 driving simulation scenario
Standard Deviation of Lane Position (feet) | Day 2
  Variability of lateral lane position during a custom STISIM3 driving simulation scenario
Standard Deviation of Lane Position (feet) | Day 4
  Variability of lateral lane position during a custom STISIM3 driving simulation scenario
Standard Deviation of Lane Position (feet) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Variability of lateral lane position during a custom STISIM3 driving simulation scenario
Standard Deviation of Lane Position (feet) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Variability of lateral lane position during a custom STISIM3 driving simulation scenario
Standard Deviation of speed (miles per hour) | Pre-injury baseline
  Variability of driving speed during a custom STISIM3 driving simulation scenario
Standard Deviation of speed (miles per hour) | Day 2
  Variability of driving speed during a custom STISIM3 driving simulation scenario
Standard Deviation of speed (miles per hour) | Day 4
  Variability of driving speed during a custom STISIM3 driving simulation scenario
Standard Deviation of speed (miles per hour) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Variability of driving speed during a custom STISIM3 driving simulation scenario
Standard Deviation of speed (miles per hour) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Variability of driving speed during a custom STISIM3 driving simulation scenario
Number of drives per day (count) | Up to 9 days post-injury
  Total number of drives per day captured as a naturalistic driving outcomes
Distance travelled per day (miles) | Up to 9 days post-injury
  Total distance driven per day captured as a naturalistic driving outcomes
Drive time per day (minutes) | Up to 9 days post-injury
  Total drive time per day captured as a naturalistic driving outcomes
Total symptom severity score | Day 2
  Total sum of 0-6 ratings across 22 symptom items (SCAT6)
Total symptom severity score | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Total sum of 0-6 ratings across 22 symptom items (SCAT6)
Total symptom severity score | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Total sum of 0-6 ratings across 22 symptom items (SCAT6)
Verbal Memory | Day 2
  Verbal memory domain score from CNS Vital Signs
Verbal Memory | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Verbal memory domain score from CNS Vital Signs
Verbal Memory | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Verbal memory domain score from CNS Vital Signs
Visual Memory | Day 2
  Visual memory domain score from CNS Vital Signs
Visual Memory | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Visual memory domain score from CNS Vital Signs
Visual Memory | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Visual memory domain score from CNS Vital Signs
Psychomotor Speed | Day 2
  Psychomotor speed domain score from CNS Vital Signs
Psychomotor Speed | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Psychomotor speed domain score from CNS Vital Signs
Psychomotor Speed | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Psychomotor speed domain score from CNS Vital Signs
Reaction Time | Day 2
  Reaction time domain score from CNS Vital Signs
Reaction Time | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Reaction time domain score from CNS Vital Signs
Reaction Time | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Reaction time domain score from CNS Vital Signs
Complex attention | Day 2
  Complex attention domain score from CNS Vital Signs
Complex attention | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Complex attention domain score from CNS Vital Signs
Complex attention | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Complex attention domain score from CNS Vital Signs
Cognitive Flexibility | Day 2
  Cognitive flexibility domain score from CNS Vital Signs
Cognitive Flexibility | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Cognitive flexibility domain score from CNS Vital Signs
Cognitive Flexibility | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Cognitive flexibility domain score from CNS Vital Signs
Processing Speed | Day 2
  Processing speed domain score from CNS Vital Signs
Processing Speed | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Processing speed domain score from CNS Vital Signs
Processing Speed | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Processing speed domain score from CNS Vital Signs
Executive function | Day 2
  Executive functions domain score from CNS Vital Signs
Executive function | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Executive functions domain score from CNS Vital Signs
Executive function | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Executive functions domain score from CNS Vital Signs
Balance Error Scoring System Total Error Score (count) | Day 2
  Number of errors committed during the Balance Error Scoring System
Balance Error Scoring System Total Error Score (count) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Number of errors committed during the Balance Error Scoring System
Balance Error Scoring System Total Error Score (count) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Number of errors committed during the Balance Error Scoring System
Tandem Gait Time (seconds) | Day 2
  Seconds to complete the tandem gait task
Tandem Gait Time (seconds) | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Seconds to complete the tandem gait task
Tandem Gait Time (seconds) | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Seconds to complete the tandem gait task
Smooth Pursuit Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Smooth Pursuit Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Smooth Pursuit Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal Saccades Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal Saccades Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal Saccades Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical Saccades Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical Saccades Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical Saccades Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Convergence Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Convergence Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Convergence Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal VOR Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal VOR Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Horizontal VOR Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical VOR Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical VOR Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Vertical VOR Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Visual Motion Sensitivity Symptom Rating | Day 2
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Visual Motion Sensitivity Symptom Rating | Within 24 hours of when symptoms resolve (Asymptomatic) (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening
Visual Motion Sensitivity Symptom Rating | Within 24 hours of unrestricted medical clearance (on average <30 days post-concussion - tracked up to 1 year)
  Sum of 0-10 ratings across 4 symptom items as part of Vestibulo-Ocular Motor Screening

SECONDARY OUTCOMES:
Pedestrian Collisions (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of pedestrian collisions during a custom STISIM3 driving simulation scenario
Speed exceedances (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of speed exceedances during a custom STISIM3 driving simulation scenario
Percent time over speed limit (%) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Percent time over speed limit during a custom STISIM3 driving simulation scenario
Percent time out of lane (%) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Percent time out of lane during a custom STISIM3 driving simulation scenario
Lateral lane position (feet) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Lateral lane position during a custom STISIM3 driving simulation scenario
Speed (miles per hour) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Driving speed during a custom STISIM3 driving simulation scenario
Number of speeding events (count) | Up to 9 days post-injury
  Number of speeding events captured as a naturalistic driving outcomes
Hard braking events (count) | Up to 9 days post-injury
  Hard braking events captured as a naturalistic driving outcomes
Hard acceleration events (count) | Up to 9 days post-injury
  Hard acceleration events captured as a naturalistic driving outcomes
Hard cornering events (count) | Up to 9 days post-injury
  Hard cornering events captured as a naturalistic driving outcomes
UFOV Processing Speed (ms) | Day 2, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Processing Speed task performance during Useful Field of View Test
UFOV Divided Attention (ms) | Day 2, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Divided attention task performance during Useful Field of View Test
UFOV Selective Attention (ms) | Day 2, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Selective attention task performance during Useful Field of View Test
Rey Osterrieth Copy Score (count) | Day 2, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Number of correct items when drawing figure during a Rey Osterrieth copy trial
Rey Osterrieth Copy Time (sec) | Day 2, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Time to draw a figure during a Rey Osterrieth copy trial

OTHER OUTCOMES:
Stop light tickets (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of stop light tickets during a custom STISIM3 driving simulation scenario
Stop sign tickets (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of stop sign tickets during a custom STISIM3 driving simulation scenario
Turn signal use (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of turn signal use during a custom STISIM3 driving simulation scenario
Tailgating (count) | Pre-injury baseline, day 2, day 4, within 24 hours of when symptoms resolve (Asymptomatic), within 24 hours of unrestricted medical clearance
  Count of tailgating events during a custom STISIM3 driving simulation scenario

CONTACTS AND LOCATIONS:
Overall Officials: Julianne Schmidt, PhD, ATC, Principal Investigator — University of Georgia
Locations (1):
- Ramsey Student Center, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided